CLINICAL TRIAL: NCT06774196
Title: Integrating Behavioral Therapy in the Management of Temporomandibular Disorders: A Comprehensive Evaluation Using DC/TMD Axis II Criteria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Khalid University (Other)
Responsible Party: Principal Investigator, Sunil Kumar Vaddamanu, Assistant Professor, King Khalid University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECM#2024-3196
Record Dates: First submitted 2025-01-02; First posted 2025-01-14 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-01

CONDITIONS: Temporomandibular Joint Disorders; Chronic Pain; Anxiety Disorders
Keywords: Temporomandibular Disorders; Temporomandibular Joint; Cognitive Behavioral Therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders; Chronic Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Therapy Group (Experimental): Participants receiving behavioral therapy (Cognitive Behavioral Therapy, relaxation techniques, and biofeedback).
  Interventions: Behavioral: Behavioral Therapy Group
- Standard Care Group (Active Comparator): Participants will receive standard care, consisting of pharmacological treatment (e.g., NSAIDs, muscle relaxants) and physical therapy.
  Interventions: Procedure: Standard Care Group

INTERVENTIONS:
Behavioral: Behavioral Therapy Group — Includes Cognitive Behavioral Therapy (CBT), relaxation techniques, and biofeedback.
  Arms: Behavioral Therapy Group
Procedure: Standard Care Group — Includes pharmacological treatment (e.g., NSAIDs, muscle relaxants) and physical therapy interventions
  Arms: Standard Care Group

SUMMARY:
This study evaluates the efficacy of behavioral therapy, including Cognitive Behavioral Therapy (CBT), relaxation techniques, and biofeedback, in managing Temporomandibular Disorders (TMD). It aims to address both the physical and psychological aspects of TMD, focusing on pain reduction, improved jaw function, and alleviating psychological distress such as anxiety and depression. Participants are randomized into two groups: an intervention group receiving behavioral therapy and a control group receiving standard care. Outcomes will be assessed using validated tools to measure pain intensity, jaw function, and psychological well-being at baseline, post-treatment, and at a 6-month follow-up. This research seeks to establish the role of behavioral therapy as a key component in the comprehensive management of TMD.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years.
* Diagnosed with Temporomandibular Disorders (TMD) based on DC/TMD Axis I and Axis II criteria.
* Presenting with symptoms such as jaw pain, limited jaw movement, or psychosocial distress (anxiety, depression).
* Willing and able to provide informed consent.
* Able to comply with the study protocol and attend all follow-up visits.

Exclusion Criteria:

* Severe systemic diseases or other neurological conditions that could interfere with treatment or outcomes.
* History of psychiatric disorders unrelated to TMD, such as schizophrenia or bipolar d disorder.
* Pregnant or lactating women.
* Use of medications or treatments within the past month that could influence study outcomes (e.g., corticosteroids, strong analgesics).
* Individuals with severe dental or maxillofacial conditions requiring immediate surgical intervention.
* Non-compliance with previous medical advice or treatment for TMD. Participants unable to understand or follow the study procedures due to language barriers or cognitive impairments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Baseline, 8 weeks post-treatment, and 6-month follow-up
  Assesses changes in self-reported pain levels with scores ranging from 0 (no pain) to 10 (worst pain)levels (0 = no pain, 10 = worst pain)
Psychological Distress (Anxiety) | Baseline, 8 weeks post-treatment, and 6-month follow-up
  Measures depression levels with a score based on the frequency and severity of symptoms.
Psychological Distress (Depression) | Baseline, 8 weeks post-treatment, and 6-month follow-up
  Measures depression levels with a score based on the frequency and severity of symptoms.

SECONDARY OUTCOMES:
Maximum Mouth Opening | Baseline, 8 weeks post-treatment, and 6-month follow-up
  Measures the maximum distance (in millimeters) between the upper and lower front teeth during maximum voluntary opening.
Jaw Range of Motion | Baseline, 8 weeks post-treatment, and 6-month follow-up
  Assesses the range of motion of the jaw through physical examination, measuring angular movement in degrees.
Pain-Related Disability | Baseline, 8 weeks post-treatment, and 6-month follow-up
  Assessed using the TMD Pain Disability Index (TDI) to evaluate the impact of pain on daily activities and quality of life
Long-Term Symptom Relief | 6-month follow-up
  Sustained improvement in pain, jaw function, and psychological distress over time, assessed using VAS, GAD-7, PHQ-9, and TDI scores.

CONTACTS AND LOCATIONS:
Locations (1):
- King Khalid University, Abhā, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) from this study will not be shared with other researchers. This decision is based on the need to protect participant privacy and confidentiality, as well as the sensitive nature of the data collected, including psychological and health-related information. Although the study results will be shared in aggregated and anonymized formats through publications and presentations, no raw or identifiable participant data will be disclosed to external parties. This approach ensures compliance with ethical guidelines and data protection regulations.